CLINICAL TRIAL: NCT04709354
Title: Clinical and Dermoscopic Evaluation of Nail Findings of Rheumatoid Arthritis, Ankylosing Spondylitis and Psoriatic Arthritis Patients and Comparison With Psoriasis Patients
Brief Title: Clinical and Dermoscopic Comparison of Rheumatoid Arthritis, Ankylosing Spondylitis and Psoriasis Patients' Nails
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 54022451-050.06.06
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis Circinata; Psoriatic Arthritis; Rheumatoid Arthritis; Spondylarthropathies; Psoriatic Nail
Keywords: Psoriasis; Psoriatic Arthritis; Psoriatic Nail; Dermoscopy
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid; Spondylarthropathies; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- rheumatoid arthritis patient: Skin and fingernail examination of newly diagnosed (diagnosed before 1 year) rheumatoid arthritis patients will be done. A detailed dermoscopic examination will be performed on the nails of these patients.
  Interventions: Diagnostic Test: Dermoscopic examination
- patients with spondylopathy: Skin and fingernail examination of newly diagnosed (diagnosed before 1 year) patient with spondylopathy will be done. A detailed dermoscopic examination will be performed on the nails of these patients.
  Interventions: Diagnostic Test: Dermoscopic examination
- psoriatic arthritis: Skin and fingernail examination of patient with psoriatic arthritis will be done. A detailed dermoscopic examination will be performed on the nails of these patients. PASI and NAPSI scores of all patients will be calculated.
  Interventions: Diagnostic Test: Dermoscopic examination
- psoriasis patients without joint involvement: Skin and fingernail examination of patient with psoriasis patients without joint involvement will be done. A detailed dermoscopic examination will be performed on the nails of these patients. PASI and NAPSI scores of all patients will be calculated.
  Interventions: Diagnostic Test: Dermoscopic examination

INTERVENTIONS:
Diagnostic Test: Dermoscopic examination — The periungual area, nail plate, subungual area of the patients' fingernails will be examined and images of the lesional nails or target nails will be recorded for comparison.

SUMMARY:
This study evaluates the fingernail findings of the rheumatoid arthritis, spondylopathy and psoriatic arthritis patient groups with the fingernails of psoriasis patients clinically and dermatoscopically and investigates the benefit of dermoscopy in the differentiation of these patients.

DETAILED DESCRIPTION:
Psoriasis is a common chronic inflammatory disease with many comorbidities. Dermatologists have a very important role in the early diagnosis of psoriatic arthritis, which is one of the most important comorbidities of psoriasis. Therefore, studies have been conducted on many factors predicting the risk of psoriatic arthritis and it has been concluded that nail involvement is closely related to psoriatic arthritis.For this reason, the importance of nail examination in the follow-up of psoriasis patients has increased significantly. Nail examination should be done carefully to predict the risk of developing psoriatic arthritis, especially at the beginning of the disease and subclinical types, and dermoscopy should be used to identify patients who may be clinically uncertain.

In addition, rheumatoid arthritis and spondylopathy patients have a lot in common with psoriatic arthritis patients.In these patients, there is no clear distinction to diagnose joint involvement, and their distinction is mostly based on the presence or absence of skin findings.Nail findings have an important place among this skin findings in the diagnosis of these patients.

Based on all these, this study questions the benefit of clinical and dermoscopic examination of nail findings in the early stages to differentiate these patients, as well as comparing the nail findings and revealing the differences and similarities.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis confirmed by dermatologist.
* Rheumatoid arthritis, ankylosing spondylitis confirmed by rheumatologist (newly diagnosed).

Exclusion Criteria:

* Unable to consent and understand
* Patients with confirmed onychomycosis
* Patients receiving biological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years with psoriasis, rheumatoid arthritis, ankylosing spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Comparation of clinical features of nails | six months
  All of patients' fingernails will be examined clinically and visible nail findings will be noted. Many findings such as onycholysis, pitting, splinter hemorrhage, nail base vascularity, leukonychia etc. will be recorded. Also, the severity of nail involvement in psoriasis patients will be measured by the NAPSI score
Comparation of dermoscopic features of nails | six months
  All of patients' fingernails will be examined by dermoscopy and nail findings will be noted. Also in particular, vascularization around the nail will be checked and images of all of the findings will be taken. Rheumatoid arthritis and spondylopathy patients with nail findings consistent with psoriasis will be enrolled.
NAPSI (Psoriasis Area and Severity index) | six months
  All psoriasis patients will be scored on their nails with NAPSI (Psoriasis Area and Severity Index) scoring system.
  The correlation of PASI and NAPSI will be examined.
PASI (Psoriasis Area and Severity Index) | six months
  Skin lesions of all psoriasis patients will be scored with the PASI (Psoriasis Area and Severity Index) system.
  The correlation of PASI and NAPSI will be examined.

SECONDARY OUTCOMES:
Demographic characteristics | through study completion, an average of 6 months
  Demographic characteristics of patients will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nahide MD Onsun, Prof, Study Director — Bezmialem University; Begüm MD Güneş, Principal Investigator — Bezmialem University
Locations (1):
- Bezmialem Vakıf Univesity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yorulmaz A, Artuz F. A study of dermoscopic features of nail psoriasis. Postepy Dermatol Alergol. 2017 Feb;34(1):28-35. doi: 10.5114/ada.2017.65618. Epub 2017 Feb 7. PMID 28286468
- [Result] Wanniang N, Navya A, Pai V, Ghodge R. Comparative Study of Clinical and Dermoscopic Features in Nail Psoriasis. Indian Dermatol Online J. 2020 Jan 13;11(1):35-40. doi: 10.4103/idoj.IDOJ_51_19. eCollection 2020 Jan-Feb. PMID 32055506
- [Result] Zabotti A, Errichetti E, Zuliani F, Quartuccio L, Sacco S, Stinco G, De Vita S. Early Psoriatic Arthritis Versus Early Seronegative Rheumatoid Arthritis: Role of Dermoscopy Combined with Ultrasonography for Differential Diagnosis. J Rheumatol. 2018 May;45(5):648-654. doi: 10.3899/jrheum.170962. Epub 2018 Feb 15. PMID 29449498